CLINICAL TRIAL: NCT00927160
Title: Evaluation of the Mobile Acute Care of the Elderly (MACE) Unit
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: 08-0272
Record Dates: First submitted 2009-06-22; First posted 2009-06-24 (Estimated); Results first posted 2013-08-14 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Model of Care for Hospitalized Older Adults
Keywords: Mobile Acute Care of the Elderly Unit; Geriatric Models of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MACE group: Elderly patients admitted to the Mobile Acute Care of the Elderly Unit.
- Usual Care group: Elderly patients admitted to the general medicine service in the hospital

SUMMARY:
The purpose of this study is to determine if a new model of care, the Mobile Acute Care of the Elderly Unit is beneficial in improving patient outcomes for elderly patients admitted to the hospital.

DETAILED DESCRIPTION:
Inpatient hospitalizations for the elderly are fraught with hazards. Hospital complications such as delirium, falls, pressure ulcers are common in the elderly. These complications may be avoidable. Patient care units specializing in geriatric care, acute care of the elderly (ACE) units, were developed and tested and had demonstrated fewer patients discharged to nursing home, and improved ability of acutely ill older patients to perform basic activities of daily living at the time of discharge (1). However, ACE unit model have not been widely disseminated because of issues of financial viability and other limitations.

Mobile Acute Care of the Elderly (MACE) unit, a new model of geriatric inpatient care, was newly developed at the Mount Sinai Hospital and has been in use since July 2007.

MACE consists of a team care providers dedicated to the care of inpatient hospitalized elderly patients. The team consists of an attending geriatrician, a geriatrics fellow, a nurse practitioner, a social worker. The potential benefits of the MACE team over a general medicine medical service include specific attention to the needs of the elderly in the inpatient setting, potential complications, the avoidance of potentially harmful medications and improved communication in transition of care. Other quality outcome measures such as length of stay, re-hospitalization rates may be affected as a result of MACE care.

The purpose of the study is to evaluate patient care using quality markers including length of stay, re-hospitalization rates, patient satisfaction of patients admitted to the Mobile Acute Care of the Elderly Unit compared to a prospectively matched and propensity score matched control group from patients admitted to general medicine service.

Description of cohort group selection methods

We aim to enroll all Mobile ACE patients who satisfy our inclusion and exclusion criteria. To match patients on the General Medical Unit with similar characteristics to the Mobile ACE patients, we will match patients according to age (within 5 years), admitting diagnosis, and their ability to ambulate independently (functional status). We aim to match each Mobile ACE patient (case group) to one general medical unit patient (control group) with these matching characteristics. In order to do so, we will establish a pool of Mobile ACE patients and a pool of general medicine patients and enroll patients into each pool if they satisfy the inclusion and exclusion criteria according to a prospective matching protocol established and validated by Charpentier et al. (2)

This matching algorithm was selected because it has been demonstrated to achieve balance across prognostic factors in trials for which randomized allocation to treatment group is not possible. The method involves prospective individual matching of patients that have already been assigned to treatment groups (in this case, Mobile ACE unit and general medical unit). The method provide a methodologically rigorous alternative for achieving balance across treatment groups, with respect to important prognostic factors, in non-randomized trials where randomization is not possible.

For patients in the Mobile ACE unit who satisfy the inclusion and exclusion criteria, we will determine if there is a matching patient in the control group pool. If so, we will enroll the patient and matched the patient to the matching patient in the control group. If there is no match in the control group pool, we will enroll the patient into the case group pool. Because we aim to match patients concurrently, we will only match patients who have admission dates within 180 days of each other.

For patients in the general medical unit who satisfy the inclusion and exclusion criteria, the matching characteristics will be assessed and if there is a match in the pool of case group patients, the patient will be enrolled. If there is no successful match in the case group patients, we will enroll the patient to the pool of control group patients if the pool of control group patients is fewer than a predetermined size of 10 patients; or if the pool of control group patients is more than 10 patients, we will enroll the patient randomly by a predetermined probability to be in the pool of control group patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to general medical service either to Mobile Acute Care of the Elderly (MACE) Unit or to general medicine 75 years or older.
* Patients or surrogates must be reachable by the phone.
* Patient must have a Sinai affiliated physician who is identified by patient or surrogate to be primary care provider

Exclusion Criteria:

* The patient is less than 75 years old.
* The patient was admitted to specialty services including cardiology-telemetry unit, intensive care, surgery, Respiratory Care Unit (RCU).
* The patient was previously admitted to an outside hospital and now transferred to Mount Sinai for further care.
* The patient cannot be contacted by telephone.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older adults hospitalized with a general medical condition in a tertiary hospital in an urban setting
Sampling Method: Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2009-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Hung, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Landefeld CS, Palmer RM, Kresevic DM, Fortinsky RH, Kowal J. A randomized trial of care in a hospital medical unit especially designed to improve the functional outcomes of acutely ill older patients. N Engl J Med. 1995 May 18;332(20):1338-44. doi: 10.1056/NEJM199505183322006. PMID 7715644
- [Background] Charpentier PA, Bogardus ST, Inouye SK. An algorithm for prospective individual matching in a non-randomized clinical trial. J Clin Epidemiol. 2001 Nov;54(11):1166-73. doi: 10.1016/s0895-4356(01)00399-7. PMID 11675169
- [Derived] Hung WW, Ross JS, Farber J, Siu AL. Evaluation of the Mobile Acute Care of the Elderly (MACE) service. JAMA Intern Med. 2013 Jun 10;173(11):990-6. doi: 10.1001/jamainternmed.2013.478. PMID 23608775

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is an observational study which enrolled patients hospitalized from November 2008 to August 2011 at the Mount Sinai Hospital from the MACE Service or general medical service.
Pre-assignment Details: No group assignment as this is observational.
Period: Overall Study
Arm/Group | MACE Group | Usual Care Group
Started | 173 | 173
Completed | 173 | 173
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MACE Group | Usual Care Group | Total
Number analyzed (Participants) | 173 | 173 | 346
Age Continuous [Mean (Standard Deviation); unit: years] | 85.2 (5.3) | 84.7 (5.4) | 85.0 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 126 | 258
  Male | 41 | 47 | 88
Region of Enrollment [Number; unit: participants]
  United States | 173 | 173 | 346

OUTCOME MEASURES:

1. Primary Outcome: Length of Hospital Stay
Time Frame: Depending on hospital stay
Measure: Mean (Standard Deviation); unit: days
Groups:
- Mobile ACE: Patients admitted to the Mobile Acute Care of the Elderly Service
- Usual Care: Matching group of patients admitted to general medical service
Arm/Group | Mobile ACE | Usual Care
Number analyzed (Participants) | 173 | 173
days | 4.6 (3.3) | 6.8 (7.6)

2. Secondary Outcome: Rehospitalization Rate
Description: 30 days for readmission rate
Time Frame: 30 days
Measure: Number; unit: percentage of particpants
Arm/Group | Mobile ACE | Usual Care
Number analyzed (Participants) | 173 | 173
percentage of particpants | 15.4 (NA) | 22.4

ADVERSE EVENTS:
Description: serious and/or other [non-serious] adverse events were not collected/assessed
Arm/Group | Mobile ACE | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes